CLINICAL TRIAL: NCT00650169
Title: Single-Dose Food In Vivo Bioequivalence Study of Clopidogrel Bisulfate Tablets (75 mg; Mylan) to Plavix® Tablets (75 mg; Bristol-Myers Squibb/Sanofi) in Healthy Volunteers
Brief Title: Food Study of Clopidogrel Bisulfate Tablets 75 mg to Plavix® Tablets 75 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CLOP-0403
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Clopidogrel

ARMS (2):
- 1 (Experimental): Clopidogrel Bisulfate Tablets 75 mg
  Interventions: Drug: Clopidogrel Bisulfate Tablets 75 mg
- 2 (Active Comparator): Plavix® Tablets 75 mg
  Interventions: Drug: Plavix® Tablets 75 mg

INTERVENTIONS:
Drug: Clopidogrel Bisulfate Tablets 75 mg — 75mg, single dose fed
  Arms: 1
Drug: Plavix® Tablets 75 mg — 75mg, single dose fed
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's clopidogrel bisulfate 75 mg tablets to Bristol-Myers Squibb/Sanofi's Plavix® 75 mg tablets following a single, oral 75 mg (1 x 75 mg) dose administered under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older. 2. Sex: Male and/or non-pregnant, non-lactating female. Women of childbearing potential must have a negative serum (Beta HCG) pregnancy test performed within 14 days prior to the start of the study and on the evening prior to each dose administration. If dosing is scheduled on Sunday or Monday, the HCG pregnancy test should be given within 48 hours prior to dosing for each study period. An additional serum (Beta HCG) pregnancy test will be performed upon completion of the study.

b. Women must practice abstinence or be using an acceptable form of contraception throughout the duration of the study. No hormonal contraceptives or hormonal replacement therapies are permitted in this study. Acceptable forms of contraception include the following:

1. intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
2. barrier methods containing or used in conjunction with a spermicidal agent, or
3. surgical sterilization c. Women will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

(1) postmenopausal with an absence of menses for at least one (1) year, or (2) bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or (3) total hysterectomy d. During the course of the study, from study screen until study exit - including the washout period, all men and women of childbearing potential must use a spermicide containing barrier method of contraception in addition to their current contraceptive method. This advice should be documented in the informed consent form.

3. Weight: At least 60 kg (132 lbs) for men and 48 kg (106 lbs) for women and all subjects within 15% of Ideal Body Weight (IBW), as referenced by the Table of "Desirable Weights of Adults" Metropolitan Life Insurance Company, 1999 (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).

4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, Hepatitis B and Hepatitis C tests, HIV test, 12-lead ECG, and urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoids, cocaine, opiate screen, phencyclidine, and methadone) performed within 14 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco products within 1 year of the start of the study.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within the 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. A positive test for any drug included in the urine drug screen.
   6. History of drug and/or alcohol abuse.
3. Medications:

   1. Use of any prescription or over-the-counter (OTC) medications within 14 days prior to the initial dose of study medication.
   2. Use of any hormonal contraceptives and hormone replacement therapy within 3 months prior to study medication dosing.
   3. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic disease.
   2. Acute illness at the time of either the pre-study medical evaluation or dosing.
   3. A positive HIV, hepatitis B, or hepatitis C test.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to clopidogrel bisulfate or any other related drugs.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.
11. Ingestion of any cruciferous vegetables (ex. broccoli, brussels sprouts, etc.) or char-broiled meats within 7 days of drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-12; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Williams, M.D., Principal Investigator — Kendle International Inc.
Locations (1):
- Kendle International Inc., Morgantown, West Virginia, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html